CLINICAL TRIAL: NCT06758492
Title: A Prospective Observational Study of Video Laryngoscopy Versus Direct Laryngoscopy for Insertion of a Thin Endotracheal Catheter for Surfactant Administration in Newborn Infants
Acronym: NEU-VODEtec
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NEU-VODEtec 01
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Distress Syndrome (Neonatal); Respiratory Distress Syndrome (RDS); Video Laryngoscopy; Surfactant
Keywords: infant, newborn; respiratory distress syndrome; surfactant; video laryngoscopy
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 600 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Video laryngoscopy used to insert thin endotracheal catheter: Video laryngoscopy used to insert thin endotracheal catheter
  Interventions: Device: Video laryngoscopy used to insert thin endotracheal catheter
- Direct laryngoscopy used to insert thin endotracheal catheter: Direct laryngoscopy used to insert thin endotracheal catheter
  Interventions: Device: Direct laryngoscopy used to insert thin endotracheal catheter

INTERVENTIONS:
Device: Video laryngoscopy used to insert thin endotracheal catheter — Video laryngoscopy used to insert thin endotracheal catheter
  Groups: Video laryngoscopy used to insert thin endotracheal catheter
Device: Direct laryngoscopy used to insert thin endotracheal catheter — Direct laryngoscopy used to insert thin endotracheal catheter
  Groups: Direct laryngoscopy used to insert thin endotracheal catheter

SUMMARY:
Many premature babies have breathing difficulty after birth and receive help with a breathing machine (nasal continuous positive airway pressure, NCPAP). Some of the babies whose breathing gets worse despite NCPAP are treated with surfactant, a medication that is given directly into their windpipe (trachea). Some of the babies who are given surfactant get it through a ventilation tube (endotracheal tube, ETT), while others get it through a thin catheter that is too small for ventilation. When doctors insert a tube or a thin catheter into the windpipe of a baby, they use an instrument called a laryngoscope, which has a light at its tip, to identify the entrance. Most often doctors look directly into the baby's mouth with a standard laryngoscope to identify the entrance to the windpipe. However, newer video laryngoscopes have a camera along with the light at their tip, which displays a picture of the entrance to the windpipe on a screen. In a study performed at one hospital, doctors inserted an ETT first time more often when they used a video laryngoscope.

The investigators are doing a study at many hospitals where doctors usually use a standard laryngoscope to insert tubes and thin catheters into a baby's trachea by looking directly into the mouth. Each hospital will switch one-by-one to using a video laryngoscope when inserting a tube. The investigators will compare the information we collect to see if more babies who have a tube inserted first time without falls in their oxygen levels or heart rate with a video laryngoscope. The investigators will also collect information on babies who have a thin catheter inserted to compare whether doctors use fewer attempts when they use a video laryngoscope.

DETAILED DESCRIPTION:
Many newborn infants have breathing difficulty after birth, particularly when they are born prematurely. Many of these infants are supported with nasal continuous positive airway pressure (NCPAP). Some of the infants deteriorate despite treatment with NCPAP and have a thin catheter inserted into their trachea for the administration of surfactant, which is then immediately removed (often referred to as "less-invasive surfactant administration" or LISA). Insertion of a thin catheter is usually performed by doctors who are experienced at intubation (i.e. inserting endotracheal tubes, ETTs). They look directly into the the infants mouth using a standard laryngoscope to identify the opening of the airway (i.e. perform direct laryngoscopy). More recently video laryngoscopes have been developed. These devices display a magnified image of the airway on a screen that can be viewed indirectly by the doctor attempting to insert the ETT or thin catheter, and also by others. A single centre study reported that more infants were successfully intubated at the first attempt when doctors performed indirect video laryngoscopy compared to direct laryngoscopy.

It is possible to independently verify when a doctor has correctly inserted and ETT, for example by detecting carbon dioxide coming out of the tube or seeing condensation in the tube during exhalation, or by hearing breath sounds by listening to the chest during positive pressure inflations. It is not possible to independently verify whether a doctor has correctly inserted a thin catheter under direct laryngoscopy, by these or other means. The standard (and to date only) way of confirming that a thin catheter has been correctly inserted is to rely on the report of the operator. Video laryngoscopy, in contrast, allows the independent verification of the tip of a thin catheter by one or more people observing the screen.

The investigators are performing NEU-VODE, a stepped wedge cluster randomised study of the introduction of video laryngoscopy versus direct laryngoscopy for the intubation of newborn infants. Alongside this study, the investigators are performing a study of infants who have a thin endotracheal catheter inserted under video laryngoscopy versus direct laryngoscopy. As it is not possible to measure the outcome of successful insertion of the thin catheter equally in both groups, this is a prospective observational cohort study. The investigators will record information on infants who have a thin catheter inserted into the trachea for the purpose of surfactant administration at centres participating in the NEU-VODE study. The type of laryngoscope used for thin catheter insertion attempts will not be mandated; instead, the investigators will compare the information of groups within the cohort who have their first attempt made using the video laryngoscope to the group who have their first attempt made with direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* newborn infants of any sex who are are having a thin catheter inserted into their trachea for the purpose of surfactant administration

Exclusion Criteria:

* no parental consent provided to share their data

Ages: 0 Minutes to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants (<28 days old) who have a thin catheter inserted into their trachea for the purpose of surfactant administration ("less-invasive surfactant administration", LISA)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful thin catheter insertion at the first attempt without physiologic instability | At 30 minutes from the start of the insertion attempt
  Successful thin catheter insertion at the first attempt without fall in SpO2 >20% from baseline or HR<100bpm

SECONDARY OUTCOMES:
Successful thin catheter insertion at the first attempt | At 30 minutes from the start of the insertion attempt
  Successful thin catheter insertion at the first attempt
Physiologic instability during first thin endotracheal catheter insertion attempt | At 30 minutes from the start of the insertion attempt
  Fall in SpO2>20% from baseline or HR<100bpm during first thin endotracheal catheter insertion attempt
Duration of laryngoscopy of first insertion attempt | At 30 minutes from the start of the insertion attempt
  Interval from introduction of laryngoscopy blade to its removal (seconds)
Number of attempts taken to insert thin endotracheal catheter | At 30 minutes from the start of the insertion attempt
  Number of attempts taken to insert thin endotracheal catheter
Time taken to insert thin endotracheal catheter on successful attempt | At 30 minutes from the start of the insertion attempt
  Interval from insertion of laryngoscope blade to insertion of thin endotracheal catheter on successful attempt (seconds)
Total laryngoscopy time to successful insertion | At 30 minutes from the start of the insertion attempt
  Sum of all intervals from introduction of laryngoscope blade to removal for unsuccessful insertion attempts; plus interval from introduction of blade to catheter insertion for successful attempt in seconds
Lowest oxygen saturation (SpO2) during the procedure | At 30 minutes from the start of the insertion attempt
  Lowest oxygen saturation (SpO2) during the procedure
Lowest heart rate (HR) during the procedure | At 30 minutes from the start of the insertion attempt
  Lowest heart rate (HR) during the procedure
Oral trauma | At 1 hour from the start of the insertion attempt
  Oral trauma reported by clinicians
Chest compressions | At 1 hour from the start of the insertion attempt
  Chest compressions
Adrenaline | At 1 hour from the start of the insertion attempt
  Adrenaline
Further thin catheter surfactant treatment | Within 72 hours of insertion attempt
  Further thin catheter surfactant treatment
Endotracheal intubation and ventilation | Within 72 hours of insertion attempt
  Endotracheal intubation and ventilation
Surfactant treatment via endotracheal tube | Within 72 hours of insertion attempt
  Surfactant treatment via endotracheal tube

CONTACTS AND LOCATIONS:
Overall Officials: Colm P.F. O'Donnell, MB PhD, Principal Investigator — National Maternity Hospital, Dublin, Ireland
Locations (16):
- Croatia (2):
  - Clinical Hospital Centre, Rijeka
  - Clinical Hospital "Holy Spirit", Zagreb
- Czechia (3):
  - University Hospital Brno, Brno
  - General University Hospital, Prague
  - Institute for Mother and Child Care, Prague
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Second Semmelweiss University, Budapest, Hungary
- University of Padova, Padua, Italy
- Oslo University Hospital, Oslo, Norway
- Poland (4):
  - Medical University of Gdańsk, Gdansk
  - Medical University of Silesia, Katowice
  - Poznań University of Medical Sciences, Poznan
  - Provincial Hospital No. 2, Rzeszów
- Romania (2):
  - Clinical County Emergency Hospital, Sibiu
  - George Emil Palade University, Târgu Mureş
- University and Polytechnic Hospital La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared o consideration of reasonable request to investigators
Time Frame: Study publication, for 2 years